CLINICAL TRIAL: NCT02662244
Title: Long-pulsed 1064 nm Nd:YAG Laser Treatment of Basal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Arisa Ortiz, Director, Laser and Cosmetic Dermatology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160062
Record Dates: First submitted 2015-01-25; First posted 2016-01-25 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yag Laser Treatment Of Basal Cell Carcinoma (Experimental): Study participants will be treated with long-pulsed 1064 nm Nd:YAG laser at the investigator's discretion based on the clinical endpoint (slight contraction and greying of the skin surface), the tumor characteristics, and the patient's skin phototype.
  Interventions: Device: Nd:YAG laser

INTERVENTIONS:
Device: Nd:YAG laser — Long-Pulsed 1064 NM ND:Yag Laser Treatment Of Basal Cell Carcinoma

SUMMARY:
Basal cell carcinoma (BCC) is the most common skin cancer worldwide. Although this tumor is rarely life threatening, it is locally destructive and can cause significant cosmetic and functional problems. Standard therapeutic modalities for BCC often result in disfigurement from surgical treatments and recurrences with topical therapies. Thus, there is a need for alternative non-surgical options that are effective, efficient, and have a low risk of side effects. This has led to the emergence of laser investigations for the treatment of BCC due to the ease of treatment, lack of significant downtime, decreased risk of complications, and absence of a surgical scar. The primary objective of this study is to evaluate the safety and efficacy of laser treatment of subjects with BCC on the trunk and extremities. Subjects will receive one treatment with the laser to the BCC. Standard excision will be performed between 30 and 90 days after laser treatment to evaluate resolution of the BCC. A visit for suture removal will be performed as appropriate for the site of the surgery. Standardized photographs and measurements will be taken at the baseline visit, immediately after laser treatment and on the day of excision.

DETAILED DESCRIPTION:
Study visits and parameters to be measured

All visits in this study will be performed at the University of California, San Diego Dermatology Clinic, 3rd floor, 8899 University Center Ln., San Diego, California 92109.

Baseline Visit and Laser exposures (Visit 1)

This visit is expected to take approximately 1 hour. The following describes the procedures performed at this visit.

1. Prior to any screening assessments, informed consent will be obtained by the investigator. When the subject fully understands the nature of the study and its risks, the subject will be asked to sign and date the informed consent form. The investigator will then sign and date the form.
2. A detailed medical history of information pertaining to treatment will be obtained.
3. The subject will be examined to determine if he or she meets the study criteria.
4. If the subject meets the criteria for the study, the subject will be assigned the next consecutive subject number.
5. Females of childbearing age will undergo a urine pregnancy test
6. Clean skin within the test sites with alcohol and shave hair with disposable shavers (if hairs are present within the test areas)
7. The lesions to be treated will be identified and marked. A record of the location of the lesion will be made. Marking will be done to include the tumor and a 4mm margin of normal skin using a surgical marking pen.
8. The treatment area will be photographed. Emphasis will be place on keeping the ambient lighting, facial expression and camera angles exactly the same for each scheduled photograph during the study. In addition, effort will be made to include anatomic landmarks.
9. The tumor will be irradiated with appropriate overlapping laser pulses with a 5-7 mm spot from the laser with the 1064nm laser with energy settings determined to be appropriate by the study investigator as described above. A 4 mm margin zone will be included.
10. The treatment area will be photographed again.
11. The treatment area will be assessed for side effects using the following scale:

    * 0 = absence
    * 1 = mild
    * 2 = moderate
    * 3 = severe
12. The subject will be instructed on post-treatment care of the treatment areas including washing the area twice daily and applying topical antibiotic, sun avoidance and sun protection. A dressing will be applied following treatment. Subjects will be encouraged to call the investigator if they experience any adverse effects that may be related to the study.

Final Evaluation Visits (Visit 2)

30 to 90 days after laser treatment, all subjects are required to return for excision of the tumor site as located and recorded at the time of the first treatment. At this final follow-up visit, there is no will be no laser treatment. The following procedures and assessments will be performed.

1. The lesional areas to be treated will be located. A record of the size of the lesional area will be made.
2. The lesional area will be photographed.
3. The treatment area will be assessed for side effects using the following scale:

   * 0 = absence
   * 1 = mild
   * 2 = moderate
   * 3 = severe
4. The lesion will be surgically excised, using standard surgical techniques, and following the original tumor margins plus 4mm as determined and recorded at the initial visit.
5. Study participant will be instructed in standard post-operative care of the surgical site. Participant will return in 2 weeks for suture removal.

Drugs to be used

No systemic drugs will be used in this study. Local injections of 1% lidocaine with epinephrine will be used at the end of the study in order to perform an excision of the basal cell carcinoma. This is standard therapy that the study subject would have undergone without participating in the study.

Devices to be used

Cutera 532/1064nm Laser

The treatment device consists of a KTP (potassium titanyl phosphate) laser at 532 nm as well as an Nd:YAG laser emitting light at 1064nm. It is an FDA approved device that enables the treatment of small superficial vessels to large vascular lesions. Only the 1064 nm wavelength will be used for this study. The 532 nm wavelength will be turned off for the purposes of this study. All study participants will be treated with parameters determined by the PI based on the characteristics of the basal cell carcinoma. The laser wavelength will be 1064nm with a spot sizes of 5-7mm with appropriate overlapping without dynamic cooling.

(For additional device description and specifications see attached device brochure provided by Cutera)

Procedures/surgical interventions

On the final visit, 30 to 90 days after the laser treatment has been performed the study participant will undergo a standard surgical excision of the lesion with 4mm margins as below:

* 4mm margins will be drawn around the lesion
* 1% Lidocaine with epinephrine will be infiltrated
* The area will be prepped with betadine in a sterile fashion
* This will be excised to the level of the subcutaneous fat with a number 15 bard-parker blade
* The tissue will be removed with sharp and blunt dissection
* The lateral margins of the resulting defect will be undermined with sharp and blunt dissection and hemostasis was achieved with electrocautery. Dog ear repair will be performed
* The deeper layers of the defect including subcutaneous fat will be approximated to reduce tension on the suture line
* Layered wound closure will be performed as appropriate for the surgical site. The wound will be cleaned with hydrogen peroxide, dried off, bacitracin ointment will be applied and the wound covered with a pressure dressing. The patient will be given detailed verbal and written instructions on post-operative care. Participant will return in 2 weeks for suture removal.

Data to be collected and when data is to be collected

Data to be collected throughout the study includes, the items listed in Table 1 (below).

Visit Type Visits 1 Final Visit Suture Removal

Clinical measurement of lesion size X X

Clinical evaluation of post treatment side effects X X

Photo documentation pre and post treatment X X

Histologic evaluation of tumor regression X

Removal of Sutures X

Table 1. Data to be collected throughout study on all subjects.

Biostatistical Analysis

Specific data variables (e.g. data collection sheets)

The primary outcome data collected during the study will include:

* Histologic complete regression of tumor.

Secondary outcome data scores and measurements will include

* Clinical side effects occurring after each treatment
* Clinical and photographic evidence of tumor regression

Study endpoints

This is a study to measure the efficacy of the Nd:YAG laser to cause complete regression of basal cell carcinoma. The number of tumors of each type (i.e. superficial low risk, nodular low risk) responding with complete regression will be determined. Complete response will be defined as no histologic evidence of disease. The number of partially responding tumors will also be determined. Partial response will be defined as a clinical reduction in surface area of the treated tumor, with histologic evidence of residual disease

Statistical methods

Long-pulsed Nd:YAG (yttrium aluminum garnet) 1064 nm laser treatment of BCC is expected to provide complete clinical and histologic clearance in approximately 90% of tumor based on a previous study.9 The number of subjects (n=50) in this study is chosen to provide statistical power of β≥0.8 to detect a complete response frequency of at least 80%. Approximately, this level of response is considered to be clinically significant.

A statistician will be enlisted to assist in statistical analysis of the results. A Kruskal-Wallis non-parametric one-way ANOVA will be performed for various parameters including width and length of the lesion and area of the lesion to determine if size affects the outcome of treatment. Clearance rates as determined by histology will be compared between treatment and established clearance rates for standard excision to determine statistical significance. All statistical tests of differences will be considered statistically significant ≤ 5%.

BCC tumors will be analyzed as a whole and then will be stratified by subtype. Stratification of the BCC subtypes will account for the variation in results, if any. If subjects have more than one lesion treated, each lesion will be counted separately.

The primary outcome of the study is histologic complete regression of tumor

The secondary outcome is

* Clinical and photographic evidence of extent of side effects occurring after each treatment
* Clinical and photographic evidence of tumor regression

V. Study Procedures

1. Study visits and parameters to be measured All visits in this study will be performed at the University of California San Diego Dermatology Clinic, 3rd floor, 8899 University Center Ln., San Diego, California 92109.

   Baseline Visit and Laser exposures (Visit 1) This visit is expected to take approximately 1 hour. The following describes the procedures performed at this visit.
   1. Prior to any screening assessments, informed consent will be obtained by the investigator. When the subject fully understands the nature of the study and its risks, the subject will be asked to sign and date the informed consent form. The investigator will then sign and date the form.
   2. A detailed medical history of information pertaining to treatment will be obtained.
   3. The subject will be examined to determine if he or she meets the study criteria.
   4. If the subject meets the criteria for the study, the subject will be assigned the next consecutive subject number.
   5. Females of childbearing age will undergo a urine pregnancy test
   6. Clean skin within the test sites with alcohol and shave hair with disposable shavers (if hairs are present within the test areas)
   7. The lesions to be treated will be identified and marked. A record of the location of the lesion will be made. Marking will be done to include the tumor and a 4mm margin of normal skin using a surgical marking pen.
   8. The treatment area will be photographed. Emphasis will be place on keeping the ambient lighting, facial expression and camera angles exactly the same for each scheduled photograph during the study. In addition, effort will be made to include anatomic landmarks.
   9. The tumor will be irradiated with appropriate overlapping laser pulses with a 5-7 mm spot from the laser with the 1064nm laser with energy settings determined to be appropriate by the study investigator as described above. A 4 mm margin zone will be included.
   10. The treatment area will be photographed again.
   11. The treatment area will be assessed for purpura, edema, erythema, scar or blistering using the following scale:

       * 0 = absence
       * 1 = mild
       * 2 = moderate
       * 3 = severe
   12. The subject will be instructed on post-treatment care of the treatment areas including washing the area twice daily and applying topical antibiotic, sun avoidance and sun protection. A dressing will be applied following treatment. Subjects will be encouraged to call the investigator if they experience any adverse effects that may be related to the study.

   Final Evaluation Visits (Visit 2)

   30 to 90 days after laser treatment, all subjects are required to return for excision of the tumor site as located and recorded at the time of the first treatment. At this final follow-up visit, there is no will be no laser treatment. The following procedures and assessments will be performed.
   1. The lesional areas to be treated will be located. A record of the size of the lesional area will be made.
   2. The lesional area will be photographed.
   3. The treatment area will be assessed for side effects using the following scale:

      * 0 = absence
      * 1 = mild
      * 2 = moderate
      * 3 = severe
   4. The lesion will be surgically excised, using standard surgical techniques, and following the original tumor margins plus 4mm as determined and recorded at the initial visit.
   5. Study participant will be instructed in standard post-operative care of the surgical site. Participant will return in 2 weeks for suture removal.
2. Drugs to be used No systemic drugs will be used in this study. Local injections of 1% lidocaine with epinephrine will be used at the end of the study in order to perform an excision of the basal cell carcinoma. This is standard therapy that the study subject would have undergone without participating in the study.
3. Devices to be used Cutera 532/1064nm Laser

   The treatment device consists of a KTP laser at 532 nm as well as an Nd:YAG laser emitting light at 1064nm. It is an FDA approved device that enables the treatment of small superficial vessels to large vascular lesions. Only the 1064 nm wavelength will be used for this study. The 532 nm wavelength will be turned off for the purposes of this study. All study participants will be treated with parameters determined by the PI based on the characteristics of the basal cell carcinoma. The laser wavelength will be 1064nm with a spot sizes of 5-7mm with appropriate overlapping without dynamic cooling.

   (For additional device description and specifications see attached device brochure provided by Cutera)
4. Procedures/surgical interventions

   On the final visit, 30 to 90 days after the laser treatment has been performed the study participant will undergo a standard surgical excision of the lesion with 4mm margins as below:
   * 4mm margins will be drawn around the lesion
   * 1% Lidocaine with epinephrine will be infiltrated
   * The area will be prepped with betadine in a sterile fashion
   * This will be excised to the level of the subcutaneous fat with a number 15 bard-parker blade
   * The tissue will be removed with sharp and blunt dissection
   * The lateral margins of the resulting defect will be undermined with sharp and blunt dissection and hemostasis was achieved with electrocautery. Dog ear repair will be performed
   * The deeper layers of the defect including subcutaneous fat will be approximated to reduce tension on the suture line
   * Layered wound closure will be performed as appropriate for the surgical site. The wound will be cleaned with hydrogen peroxide, dried off, bacitracin ointment will be applied and the wound covered with a pressure dressing. The patient will be given detailed verbal and written instructions on post-operative care. Participant will return in 2 weeks for suture removal.
5. Data to be collected and when data is to be collected Data to be collected throughout the study includes, the items listed in Table 1 (below).

Visit Type Visits 1 Final Visit Suture Removal

Clinical measurement of lesion size X X

Clinical evaluation of post treatment side effects X X

Photo documentation pre and post treatment X X

Histologic evaluation of tumor regression X

Removal of Sutures X

Table 1. Data to be collected throughout study on all subjects.

VI. Biostatistical Analysis

1. Specific data variables (e.g. data collection sheets)

   The primary outcome data collected during the study will include:
   * Histologic complete regression of tumor Secondary outcome data scores and measurements will include
   * Clinical and photographic evidence of extent of side effects occurring after each treatment
   * Clinical and photographic evidence of tumor regression
2. Study endpoints This is a study to assess the efficacy of the Nd:YAG laser to cause complete regression of basal cell carcinoma. The number of tumors of each type (i.e. superficial low risk, nodular low risk) responding with complete regression will be determined. Complete response will be defined as no histologic evidence of disease. The number of partially responding tumors will also be determined. Partial response will be defined as a clinical reduction in surface area of the treated tumor, with histologic evidence of residual disease
3. Statistical methods Long-pulsed Nd:YAG 1064 nm laser treatment of BCC is expected to provide complete clinical and histologic clearance in approximately 90% of tumor based on a previous study.9 The number of subjects (n=50) in this study is chosen to provide statistical power of β≥0.8 to detect a complete response frequency of at least 80%. Approximately, this level of response is considered to be clinically significant.

A statistician will be enlisted to assist in statistical analysis of the results. A Kruskal-Wallis non-parametric one-way ANOVA will be performed for various parameters including width and length of the lesion and area of the lesion to determine if size affects the outcome of treatment. Clearance rates as determined by histology will be compared between treatment and established clearance rates for standard excision to determine statistical significance. All statistical tests of differences will be considered statistically significant ≤ 5%.

BCC tumors will be analyzed as a whole and then will be stratified by subtype. Stratification of the BCC subtypes will account for the variation in results, if any. If subjects have more than one lesion treated, each lesion will be counted separately.

The primary outcome of the study is histologic complete regression of tumor . The secondary outcome is clinical and photographic evidence of extent of side effects occurring after each treatment

* Clinical and photographic evidence of tumor regression

VII. Risks and Discomforts

1. Complications of surgical and non surgical procedures The laser device will be used under the immediate direction of the principal investigator and co-investigator, Drs. Arisa Ortiz and Brian Jiang, who are laser certified operator. Only credentialed laser users at the hospital can operate the device. Only Dr. Ortiz and Jiang will operate the device. Dr. Ortiz will report any minor or major adverse events (per the University of California HRPP (Human Research Protections Program) reporting guidelines that occur during the study, immediately to the UCSD Human Research Protections Program. Any risk of eye damage in subjects participating in this study will be eliminated by the wearing of protective eyewear during laser use.

   Laser pulses will produce an immediate sensation comparable to a pin-prick or rubber band snapping against the skin (mild to moderate pain) at the treatment site, and there may be a transient sensation of sunburn after irradiation that disappears over a period of several days. The following is a list of potential adverse events that could occur from use of the laser device in this study. Please note that the goal of the laser therapy is to produce damage and necrosis to the tumor. Therefore signs of this effect, including inflammation and purpura are expected outcomes and will not be recorded as adverse events.

   Subjects enrolled may expect some side effects (purpura, erythema, and edema) at the laser-treated site. Erythema and edema usually disappear within 24 to 72 hours. Purpura may persist for approximately one to two weeks. Blistering and scaling at the treated sites may also develop but are rare and temporary. Scarring, ulceration, post-inflammatory hyperpigmentation or hypopigmentation, and infection also occur rarely. The risk of infection will be minimized by proper wound care. If infection is evident at the treated site at the time of scheduled excision, the infection will be treated appropriately and the excision will be postponed for up to 2 weeks until the infection is resolved.

   Standard excision for BCC is associated with a small risk of recurrence. This risk is not increased as a result of the study.

   Subjects will be provided post laser-treatment and post excision instructions (see attached).
2. Drug side effects and toxicities The only drug used in this protocol is lidocaine/epinephrine for local anesthesia. Patients will be asked regarding allergy to medications. No adverse effect is anticipated. However, allergic reaction may occur with any medication.
3. Device complications/malfunctions Laser device Operating or treating with the device is restricted to authorized and trained personal. If the investigator has any evidence of a device malfunction that is potentially hazardous for the subject or is interfering with the performance of the device, the treatment shall be immediately interrupted and the IRB will be notified.

   Eye injury due to use of the laser system is a risk to the subject and the operator. Goggles will be labeled for specific use with the 1064 nm laser. Subjects and investigators and anyone present in the room will wear appropriate protective goggles during the procedure to avoid potential eye injury.
4. Psychosocial (non-medical) risks The investigators do not anticipate any psychosocial risks due to this study. However if any participants experience emotional distress during the study the investigators will assist them to resolve this stress with appropriate referrals. Steps to prevent this outcome will include detailed explanation of the study and what to expect from the study treatment.
5. Radiation risks This laser does not emit any ionizing radiation. Therefore, the risk associated with this type of radiation is non-existent. This laser emits light only in the visible and infrared range of the optical spectrum and therefore only thermal interaction with the tissue can be expected.

VIII. Potential Benefits

1. Potential benefits to participating individuals There will be no direct benefit to the subjects participating in the study
2. Potential benefits to society The results of this study will help us acquire information that may lead to the development of an improved treatment for skin cancer.

X. Monitoring and Quality Assurance

1. Independent monitoring of source data

   At this time the investigators do not anticipate a need for an independent monitor as our monitoring of the data will be sufficient to ensure the validity and integrity of the data and adherence to the IRB-approved protocol.

   Patients will be recruited during their scheduled office visit in the exam room. Consent will be obtained in the exam room, where patients will have the opportunity to ask the physician questions.

   The investigators will make every effort to accurately document all data on study case report forms. All source data will be organized and filed into individual subject binders. Any pertinent notes to file regarding the subject shall be documented by a study investigator and kept in the applicable subject binder. The principal investigator shall review data on an ongoing and consistent basis throughout the duration of the study. Study numbers will be used to deidentify patients. All subjects must be assigned a study identification number that is the only item that appears on the subject binder and photographs. Electronic digital images, labeled with the study identification number, will be stored both in the patient binders and on a secured hospital server. Only investigators involved in the study will have access to this data. Even with these precautions, there is a risk of loss of confidentiality. If this occurs, the subject will be notified immediately.

   This study shall be performed in accordance with all applicable federal, state and local laws and regulations, including without limitation 21 CFR Parts 50 and 56 and the Health Insurance portability and Accountability Act of 1996 ("HIPAA") and any regulations and official guidance promulgated there under.
2. Safety monitoring Safety data will be collected at each visit of the study. Investigators will perform overall efficacy assessments of this study. The Principal Investigator will be reviewing data on an ongoing and consistent basis throughout the duration of the study. The Principal Investigator is responsible for protecting the rights, safety, and welfare of subjects under his/her care. The Principal Investigator will be responsible for this review and for determining whether the research should be altered or stopped. If any severe adverse effect or death directly related to the procedure proposed occurs, Principal Investigator will report to the IRB.
3. Outcomes monitoring Any adverse events will be reviewed and analyzed by the Principal Investigator as soon as the event occurs and will be documented in the subject's binder. Any unexpected adverse reactions will be reported by telephone to the IRB within 48 hours of observing the event. If a unexpected side effect occurs, Principal Investigator will also report adverse events to the FDA.
4. Adverse event reporting guidelines The principal investigator will follow the UCSD Human Research Committee guidelines for Adverse Event Reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven basal cell carcinoma of any non-aggressive subtype less than 2 cm located on the trunk (chest, abdomen, back) or extremities (arms, legs), with clearly visible margins, suitable for treatment by standard surgical excision.
2. Age greater than 18 years.
3. Able to read and comprehend the informed consent form.
4. Informed consent form signed by the subject.
5. Willingness to follow the treatment schedule and post treatment care requirement.

Exclusion Criteria:

1. Lesion to be treated is on the face, areola, hands, feet, ankles, pretibial surface or genitalia.
2. BCC with aggressive features including morpheaform/fibrosing/sclerosing, infiltrating, perineural, metatypical/keratotic, micronodular, or basosquamous subtypes.
3. Any BCC lesion that falls under Mohs Micrographic Surgery Appropriate Use Criteria for lesions on the trunk or extremities including recurrent lesions, aggressive subtypes, tumors > 2 cm, lesions on the hands, feet, ankles, genitalia, and pretibial surface)
4. Confluent carcinomatosis in which collision lesions are likely and tumor borders are difficult to ascertain.
5. Scarring or infection of the area to be treated
6. Subject is pregnant.
7. Subject is immunocompromised. Immunocompromised is defined by any condition, process or medication that causes the immune system to be attenuated. (ie. HIV, immunosuppressive medications, active systemic malignancies, organ transplant recipients, etc).
8. Subjects with Gorlin's syndrome (Basal Cell Nevus Syndrome) or other syndrome that increases the risk of confluent carcinomatosis
9. Subjects may not be on any blood thinners, including but not limited to warfarin or clopidogrel (NOT including aspirin).
10. Prisoners and decisionally impaired subjects.
11. Current or history of psychiatric disease, or substance abuse that would interfere with ability to comply with the study protocol or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arisa Ortiz, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-three subjects seeking treatment for biopsy-proven BCC that did not meet the criteria for Mohs surgery were recruited from the clinic
Groups:
- All Participants: Subjects received one treatment with the 1064 nm Nd:YAG laser as follows: 5-6 mm spot, fluence of 125-140 J/cm2 and a pulse duration of 7-10 ms. Standard excision with 5 mm clinical margins was performed at 30 days after laser treatment to evaluate clinical and histologic clearance of BCC.
Period: Overall Study
Arm/Group | All Participants
Started | 33
Completed | 31
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Yag Laser Treatment Of Basal Cell Carcinoma: Thirty-one subjects seeking treatment for biopsy-proven BCC that did not meet the criteria for Mohs surgery were recruited. Subjects on current anticoagulation therapy, or with a history of immunosuppression were excluded. Subjects received one treatment with the 1064 nm Nd:YAG laser as follows: 5-6 mm spot, fluence of 125-140 J/cm2 and a pulse duration of 7-10 ms. Standard excision with 5 mm clinical margins was performed at 30 days after laser treatment to evaluate clinical and histologic clearance of BCC. Standardized photographs and adverse assessments were taken at the baseline visit, immediately after laser treatment and on the day of excision.
  Nd:YAG laser: Long-Pulsed 1064 NM ND:Yag Laser Treatment Of Basal Cell Carcinoma
Arm/Group | Yag Laser Treatment Of Basal Cell Carcinoma
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 56 [35 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: This is a Study to Measure the Efficacy of the Nd:YAG Laser to Cause Complete Regression of Basal Cell Carcinoma.
Description: The primary outcome data collected during the study will include:
  * Number of tumors that showed histologic complete regression.
Time Frame: The primary outcome of the study is histologic clearance of BCC tumor 30 days
Population: 31 Adults over 18 years with a biopsy-proven BCC of any non-aggressive subtype with a residual clinical lesion were included. BCC lesions were required to be less than 2.1 cm in diameter and located on the trunk or extremities. The number of tumors that showed complete regression were analyzed for primary outcome.
Measure: Number; unit: tumors
Units Other Than Participants: tumors
Groups:
- Single Arm: Study participants will be treated with long-pulsed 1064 nm Nd:YAG laser at the investigator's discretion based on the clinical endpoint (slight contraction and greying of the skin surface), the tumor characteristics, and the patient's skin phototype.
  Nd:YAG laser: Long-Pulsed 1064 NM ND:Yag Laser Treatment Of Basal Cell Carcinoma
Arm/Group | Single Arm
Number analyzed (Participants) | 31
Number analyzed (tumors) | 31
tumors | 28

2. Secondary Outcome: • Clinical and Photographic Evidence of Extent of Purpura After Each Treatment
Description: 11. The treatment area will be assessed post laser and at the final evaluation visit for purpura using the following scale:
  * 0 = absence
  * 1 = mild
  * 2 = moderate
  * 3 = severe
Time Frame: 30 days
Population: All participants' purpura was analyzed on a scale of 0 to 3
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: purpura
Arm/Group | All Participants
Number analyzed (Participants) | 31
Number analyzed (purpura) | 31
score on a scale
  post baseline (5 minutes) | 0.523809524 [0 to 3]
  final visit (30 days) | 0 [0 to 3]

3. Secondary Outcome: • Clinical and Photographic Evidence of Extent of Edema Occurring After Each Treatment
Description: 3. The treatment area will be assessed for edema using the following scale:
  * 0 = absence
  * 1 = mild
  * 2 = moderate
  * 3 = severe
Time Frame: 30 days
Population: Clinical and photographic evidence of extent of edema was evaluated by the investigator with the above scores at b
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: edema
Groups:
- All Participants: Subjects received one treatment with the 1064 nm Nd:YAG laser as follows: 5-6 mm spot, fluence of 125-140 J/cm2 and a pulse duration of 7-10 ms. Standard excision with 5 mm clinical margins was performed at 30 days after laser treatment to evaluate clinical and histologic clearance of BCC.
  30 to 90 days after laser treatment, all subjects are required to return for excision of the tumor site as located and recorded at the time of the first treatment. At this final follow-up visit, there is no will be no laser treatment. The following procedures and assessments will be performed.
  1. The lesional areas to be treated will be located. A record of the size of the lesional area will be made.
  2. The lesional area will be photographed.
  3. The treatment area will be assessed for purpura, edema, erythema, scar or blistering using the following scale:
     * 0 = absence
     * 1 = mild
     * 2 = moderate
     * 3 = severe
Arm/Group | All Participants
Number analyzed (Participants) | 31
Number analyzed (edema) | 31
score on a scale
  post baseline treatment (5 minutes) | 1.428571429 [0 to 3]
  final visit (30 days) | 0 [0 to 3]

4. Secondary Outcome: Clinical and Photographic Evidence of Extent of Erythema Occurring After Each Treatment
Description: The treatment area will be assessed for erythema using the following scale:
  * 0 = absence
  * 1 = mild
  * 2 = moderate
  * 3 = severe
Time Frame: 30 days
Population: Clinical and photographic evidence of extent of erythema was evaluated by the investigator with the above scores.
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: erythema
Arm/Group | All Participants
Number analyzed (Participants) | 31
Number analyzed (erythema) | 31
score on a scale
  post baseline treatment (5 minutes) | 1.571428571 [0 to 3]
  final visit (30 days) | 1.095238095 [0 to 3]

5. Secondary Outcome: Clinical and Photographic Evidence of Extent of Blistering Occurring After Each Treatment
Description: The treatment area will be assessed for blistering using the following scale:
  * 0 = absence
  * 1 = mild
  * 2 = moderate
  * 3 = severe
Time Frame: 30 days
Population: Clinical and photographic evidence of extent of blistering after treatment was evaluated by the investigator with the above scores
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: blistering
Arm/Group | All Participants
Number analyzed (Participants) | 31
Number analyzed (blistering) | 31
score on a scale
  post baseline treatment (5 minutes) | 1.19047619 [0 to 3]
  final visit (30 days) | 0.047619048 [0 to 3]

ADVERSE EVENTS:
Description: Laser pulses will produce an immediate sensation comparable to a pin-prick or rubber band snapping against the skin (mild to moderate pain) at the treatment site, and there may be a transient sensation of sunburn after irradiation that disappears over a period of several days. All effects of laser are localized reactions like erythema, purpura, scabbing, localized hypo, hyperpigmentation. Risk of mortality cannot be expected from localized treatment.
Groups:
- Yag Laser Treatment Of Basal Cell Carcinoma: Single arm/group study
  Study participants will be treated with a long-pulsed 1064 nm Nd:YAG laser with a 5-7 mm spot, an approximate fluence of 100-200 J/cm2 and a pulse duration of 3-15ms determined somewhat at the investigator's discretion based on the clinical endpoint (slight contraction and greying of the skin surface), the tumor characteristics, and the patient's skin phototype. There will be no randomization.
Arm/Group | Yag Laser Treatment Of Basal Cell Carcinoma
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 1/31
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yag Laser Treatment Of Basal Cell Carcinoma (N=31)
pain (Skin and subcutaneous tissue disorders) | 1 (1) — pain at laser site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No